CLINICAL TRIAL: NCT06932679
Title: Affordances and Impairments: A Paradigm for Understanding Obstacle Crossing in Parkinson's Disease
Brief Title: Perception of Affordances and Obstacle Crossing in People With Parkinson's Disease and Healthy Adults
Status: Recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: University of Haifa, Israel (Unknown)
Responsible Party: Principal Investigator, Galit Yogev-Seligmann, Senior Lecturer, Department of Occupational Therapy, Faculty of Social Welfare and Health Sciences, University of Haifa, University of Haifa
Other Study IDs: 1561/25
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease; Obstacle Crossing; Gait; Affordances; Motor Control; Balance; Fall Risk; Visual Exploration; Gaze Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's Disease: Participants diagnosed with Parkinson's disease (PwP), aged 60-80 years, able to walk independently outdoors.
  Interventions: Other: Assessment of Gait and Visual Exploration
- Healthy Older Adults: Healthy adults aged 60-80 years, without neurological or orthopedic conditions affecting gait.
  Interventions: Other: Assessment of Gait and Visual Exploration
- Healthy Young Adults: Healthy adults aged 20-30 years, without neurological or orthopedic conditions affecting gait.
  Interventions: Other: Assessment of Gait and Visual Exploration

INTERVENTIONS:
Other: Assessment of Gait and Visual Exploration — Participants will perform walking tasks involving obstacle crossing while their gait and visual exploration patterns are recorded using wearable sensors and eye-tracking glasses. This is a non-invasive observational study with no therapeutic intervention.

SUMMARY:
This study aims to explore how young adults, older adults and people with Parkinson's disease (PwP), perceive their abilty to cross obstacles while walking, and how this perception is related to their actual performance of obstacle crossing and disease-related motor and cognitive impairments. The study will explore this percepeption and the actual performance in different walking environments(floor, synthetic grass turf). Understanding how people perceive obstacles may help improve rehabilitation methods and reduce the risk of falls. The study will take place at the Motor Performance Laboratory, University of Haifa, and will include walking tasks, eye-tracking measurements, and motor and cognitive assessments.

DETAILED DESCRIPTION:
This study investigates the role of affordance perception - the ability to perceive opportunities for action - during obstacle crossing in people with Parkinson's disease (PwP). Falls are highly prevalent in PwP, often resulting from tripping over obstacles. While previous research has mainly focused on gait impairments, this study uniquely examines the perceptual stage that precedes movement and the association between perception, cognition, and motor performance.

Participants will include 60 PwP and 120 healthy adults (60 older adults and 60 young adults). All participants will perform walking tasks involving obstacle crossing under different environmental conditions (e.g., different obstacle heights and surfaces). Prior to walking, participants will judge whether they can safely cross the obstacle. Eye-tracking glasses will measure visual exploration patterns to assess how participants scan the environment. Additionally, walking variables such as speed and step length, will be recorded using wearable sensors.

The study will explore:

1. Differences in affordance perception between PwP and healthy adults.
2. Associations between motor and cognitive impairments and affordance perception in PwP.
3. How affordance perception relates to gait performance during obstacle crossing.

Results from this study may help to develop new intervention strategies aimed at improving safe walking and obstacle negotiation in PwP.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 20 to 80 years.
* Ability to walk independently outdoors without assistive devices.
* For Parkinson's Disease (PD) group: Diagnosis of PD confirmed by medical records.
* For healthy control groups: No neurological or orthopedic conditions affecting gait.

Exclusion Criteria:

* Feezing of gait (for PD group only), based on a score greater than 0 on the Freezing of Gait Questionnaire.
* Severe visual impairment that cannot be corrected with glasses or lenses.
* Cognitive impairment, defined as a score below 18 on the telephone-based Mini-Mental State Examination (MMSE).
* Any orthopedic condition, pain, or other medical condition that may affect walking, based on self-report.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include three groups: (1) people with Parkinson's disease (PwP), aged 60-80 years, diagnosed by a physician and able to walk independently outdoors; (2) healthy older adults aged 60-80 years without neurological or orthopedic conditions affecting gait; and (3) healthy young adults aged 20-30 years without neurological or orthopedic conditions affecting gait.
  Participants will be recruited from the community, from clinical settings (for PwP), and through university-based recruitment systems (for young healthy adults).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2028-04-24 (Estimated); Study Completion 2028-06-24 (Estimated)

PRIMARY OUTCOMES:
Affordance Perception Accuracy | During single laboratory session (about 3 hours)
  Accuracy of participants' perception of their ability to cross obstacles of varying height and surface conditions. Participants will judge whether they can safely cross an obstacle prior to walking.
Affordances measured by gaze behavior | During a single laboratory session (approximately 3 hours)
  Eye movement patterns during obstacle approach and crossing. Gaze behavior will be recorded using wearable eye-tracking glasses (Tobii Pro Glasses 3) to assess visual exploration of the walking environment and obstacle. Measures will include fixation(on obstacle) duration (milisecondes).

SECONDARY OUTCOMES:
Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | During a single laboratory session (approximately 3 hours)
  Disease severity will be assessed using the MDS-UPDRS (Motor Examination). This standardized clinical assessment measures motor symptoms in people with Parkinson's disease, including tremor, rigidity, bradykinesia, and postural stability. Higher scores indicate greater motor impairment.
Walking Speed | During a single laboratory session (approximately 3 hours)
  Walking speed during obstacle crossing tasks, measured using wearable sensors (APDM Mobility Lab). Walking speed will be calculated in meters per second based on time and distance walked during the trials.
Step Length | During a single laboratory session (approximately 3 hours)
  Step length during obstacle crossing tasks, measured using wearable sensors (APDM Mobility Lab). Step length will be calculated in meters for each leg during walking trials, as an indicator of gait characteristics and stability.
Levodopa Equivalent Daily Dose (LEDD) | During a single laboratory session (approximately 3 hours)
  The total daily dose of antiparkinsonian medications will be calculated for participants with Parkinson's disease using the standardized Levodopa Equivalent Daily Dose (LEDD) formula. Higher values indicate greater medication use.
Cognitive Performance - Stroop Test (NeuroTrax Cognitive Battery) | During a single laboratory session (approximately 3 hours)
  Cognitive function will be assessed using the computerized NeuroTrax Cognitive Battery. Specifically, performance on the Stroop test will be used to evaluate executive function, focusing on response inhibition and attention control. The Stroop test provides accuracy and reaction time scores, with higher scores reflecting better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yogev Seligmann, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Motor Performance Laboratory, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Data collected in this study will only be used by the study investigators for research purposes, in accordance with the approved study protocol and ethical guidelines.